CLINICAL TRIAL: NCT04257734
Title: Epidemiologic and Clinical Characteristics of Optic Neuritis in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Peking University Health Science Center (Other)
Responsible Party: Principal Investigator, Wei Shihui, Professor, Chinese PLA General Hospital
Other Study IDs: CONSG1
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Optic Neuritis
Keywords: optic neuritis; clinical Characteristics; epidemiology
MeSH Terms: conditions — Optic Neuritis | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- optic neuritis: Aquaporin 4 antibody seropositive optic neuritis patients, Myelin oligodendrocyte glycoprotein antibody seropositive optic neuritis patients, and double antibodies seronegative optic neuritis patients
  Interventions: Other: observation

INTERVENTIONS:
Other: observation — different serum antibodies status

SUMMARY:
This will be a hospital-based retrospective multi-center study on epidemiologic and clinical characteristics of optic neuritis among Chinese. The investigation will cover about 29 provinces or municipalities all around China.

DETAILED DESCRIPTION:
This national investigation will be conducted to describe the epidemiology and clinical characteristics of optic neuritis in China. All the patients will be divided into 3 groups according to the serum demyelinating antibodies (Aquaporin-4 antibody seropositive group, Myelin oligodendrocyte glycoprotein antibody seropositive group and double seronegative group). The investigator will analyze the differences among the three groups.

Primary outcomes:

* To dig out the different visual acuity (VA, LogMAR) prognosis among the three groups;

  * To calculate the annual relapse rate (ARR) differences among the three groups (relapse times in all the follow-up time in each group/ follow-up time (years) in all in each group).

Secondary outcomes:

* Other epidemiological and clinical characteristics of optic neuritis patients will be analyzed among the three groups;

  * Orbital or Brain MRI is required in this study, which could avoid the misdiagnosis. We will collect and analyze these MRI data too (including the optic nerve lesions in T2 weight images and T1 enhanced MRI);

    * Results of optical coherence tomography (OCT) (including peripapillary retinal nerve fiber layer, macular thickness ,and ganglion cell and inner plexiform layer complex) at different time point are also needed in this study. However, OCT is not necessarily required;

      * Visual fields at different time points are also encouraged to provide if they are available.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of optic neuritis
2. The patients' medical records were complete

Exclusion Criteria:

1. Patients with unclear diagnosis of optic neuritis
2. Incomplete medical records

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Optic neuritis patients with complete medical records in multicenter from China.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Visual Acuity | At least 1 year from the attack to the final visit
  Last visual acuity records in the hospital
Annual Relapse Rate | At least 1 year from the attack to the final visit
  Calculated annual relapse rate of different subgroups in the cohort

SECONDARY OUTCOMES:
Epidemiologic characteristics of optic neuritis | At least 1 year from the attack to the final visit
  Gender, age of first attack, location
Clinical characteristics of optic neuritis | At least 1 year from the attack to the final visit
  Visual acuity at nadir, pain, optic disc edema
Optical Coherence Tomography | At least 1 year from the attack to the final visit
  RNFL, macular thickness and GCIPL at different time points
Orbit or Brain MRI at the attack | At least 1 year from the attack to the final visit
  Lesions of the optic nerve

CONTACTS AND LOCATIONS:
Overall Officials: Shihui Wei, M.D, Study Chair — Ophthalmology, the Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
It is a multi center study of optic neuritis, the individual participant data belongs to every single center. Now, we are applying for the approval. However, the details will not be available until all the centers approved.